CLINICAL TRIAL: NCT05181644
Title: Perspective, Randomized Controlled Study Aimed at Evaluating the Effectiveness of the EmoLED Medical Device in the Healing of Digital Ulcers in Patients Affected by Scleroderma. (S.U.I.T.A.B.L.E.)
Brief Title: Effectiveness of the EmoLED Medical Device in the Healing of Digital Ulcers in Patients With Scleroderma.
Acronym: SUITABLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to reach the expected number of patients
Sponsor: Emoled (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmoLED_004
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Ulcer; Acral Nevus; Scleroderma; Digital Ulcer
Keywords: ulcer; acral; scleroderma; EmoLED; wound healing; blue light; digital ulcer
MeSH Terms: conditions — Ulcer; Scleroderma, Diffuse; digital ulcers

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled study. It is a 1:1 randomization, stratified, with 3 blocks of patients distributed in the two groups (experimental and control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): To the Control Group is administered the current standard therapy for 16 weeks.
  Interventions: Procedure: current Standard of Care
- EmoLED Group (Experimental): The treatment with EmoLED will be carried out once a week in correspondence with the dressing change of the lesion, for sixteen consecutive weeks, for a total of 16 treatments.
  Interventions: Device: EmoLED treatment; Procedure: current Standard of Care

INTERVENTIONS:
Device: EmoLED treatment — Treatment with the EmoLED device consists of irradiating each area of 5 cm in diameter of the lesion for 60 seconds; if the lesion is larger than 5 cm in diameter, the applications will be repeated up to cover the entire area of interest. EmoLED treatment is additional to the standard therapy for the patient.
  Arms: EmoLED Group
Procedure: current Standard of Care — The acral lesions will be cleansed with physiological solution, disinfected with a special device and, if necessary, a debridement will be carried out with the most appropriate method.

SUMMARY:
The present clinical study aims to compare, in the two groups of patients with acral ulcers, the reparative process of the injured area, the evaluation of the healing time (with "healing" interpreted as the complete re-epithelization of the wound) and the perception of pain through NRS scale.

DETAILED DESCRIPTION:
This clinical study will be a prospective, randomized controlled study, with the commercial objective of assessing the clinical effectiveness of a portable battery powered device that uses blue LED.

This clinical study aims to compare the existing standard treatment for acral ulcers in patients suffering from scleroderma, to a protocol that provides for the administration of the EmoLED treatment for 16 consecutive weeks in addition to the conventional therapy.

The objective is to determine any differences in outcome between the two groups considered and whether the therapy of the treatment group is a valid alternative to the current therapy in terms of support for the reparative process, speed of healing and pain reduction.

The study protocol also establishes a follow-up period of 4 weeks. If the injury has not healed within the 16 weeks of treatment, the patient will return to the investigator centre for the usual dressing, and the evolution of the injury will be observed for 4 weeks. If the recovery occurs within the 16 weeks of treatment, the patient will return to the investigator centre 4 weeks after recovery, for a check-up, during which the condition of the healed skin area and the presence of any relapses will be evaluated.

In this clinical study, patients with systemic sclerosis with at least one ulcerative lesion on the upper limbs' fingers will be enrolled. In case the patient has more than one lesion, only one will be selected for the study; it will be the one that, in the opinion of the doctor, allows a better recording of data (image acquisition).

The population subject matter of the study is largely representative of the target population, as there are no particular exclusion criteria and the center involved is a structure of excellence in the treatment of acral ulcers of sclerodermal origin.

Scleroderma, or systemic sclerosis, is a chronic systemic disease with autoimmune pathogenesis, characterized by skin and internal organs fibrosis caused by an altered functionality of fibroblasts, the presence of perivascular inflammatory infiltration and small vessel alterations and immune system abnormalities.

The incidence of scleroderma is estimated in about twenty cases per million inhabitants per year. The peak age range for the onset of this disease is between 45 and 65 years and, as often observed in autoimmune diseases, women are more frequently affected with a ratio of 4.5:1.

Scleroderma begins in most cases with the Raynaud's phenomenon, consisting in the change of colour of the extremities, which become initially pale, then cyanotic and finally red.

The most characteristic sign of scleroderma is the thickening of the skin, that can be found at the level of the hands, which can meet a progressive deformity in fingers bending, and then also at the level of the wrists, forearms, face and trunk.

There are still no drugs that can cure scleroderma. The treatments used, therefore, aim to contain the symptoms and to avoid/delay the complications of the disease. The most commonly used drugs include vasodilators, pro-kinetic drugs, antiarrhythmics and immunosuppressants to treat the various complications.

Digital ulcers represent a complication that affects about half of patients with systemic sclerosis. Digital ulcers are mainly the consequence of vascular phenomena typical of the disease (Raynaud phenomenon and endothelial damage) or of its fibrotic evolution (skin sclerosis). They are mainly located at the extremities where peripheral vascular phenomena are more evident, at the level of the areas where the skin is most subjected to traction (e.g. the elbows), or in the areas affected by calcinosis. Ulcerations of the knuckles and fingertips are frequent.

Digital ulcers often develop a chronic trend over time, they have a slow healing, they are intensely painful and can lead to a severe functional limitation, compromising the personal and professional quality of life of the affected person, so much so that it represents one of the most important complications from this point of view, perceived by patients as seriously disabling. This type of ulcers can also lead to infectious complications (osteomyelitis, sepsis of the surrounding soft tissues) that in the most serious cases lead to the necrosis of the local tissue resulting in the amputation of the digital phalanges.

Factors to consider in assessing the type of the ulcer include location and size, margins and edges, wound bed, degree of moisture (exudate), edema (local or diffused), pain assessment and degree of infection. From these factors we can distinguish three types of ulcers: superficial, intermediate and deep. The management of a digital ulcer is particularly complex and may involve a local therapy, a systemic therapeutic approach, or a combined therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from systemic sclerosis with at least an ulcerative lesion on the fingers of the upper limbs;
* The ulcer must not present bone or tendon exposure;
* Chronicity of the lesion: at least 4 weeks;
* Men and women aged ≥ 18 years;
* The patient must be able to understand the purposes of the clinical trial and provide informed consent in writing.

Exclusion Criteria:

* Patients who are participating in other clinical trials with drug or medical device;
* Patients with a history of self-harm who can voluntarily alter the course of healing;
* Women who are pregnant or breastfeeding1;
* Patients who participated in a clinical study on the healing of skin ulcers during the previous month;
* Patients who are unable to understand the purposes and objectives of the study;
* Presence of infectious signs according to IDSA criteria at the time of recruitment;
* Presence of peripheral vascular obstructive diseases;
* Patients with psychiatric disorders;
* Patients with neoplasia;
* Patients with pathologies that induce skin photosensitivity;
* Patients with a limited life expectancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Number of healed lesions in the two groups | 16 weeks
  The primary endpoint is the comparison of the outcomes in terms of number of patients with an acral lesion that reach healing (interpreted as the complete re-epitelization of the lesioned area) treated with the standard method (Control Group), versus the number of patients with an acral lesion treated with Emoled and the standard method (Treated Group), at the last visit of the sixteen weeks of observation.

SECONDARY OUTCOMES:
Healing time evaluation | 20 weeks
  Average healing time (where "healing" means the complete re-epithelization of the observed area) during the overall weeks of observation in the two treatment groups.
Pain evaluation | 16 weeks
  Percentage of variation of perceived pain in both treatment groups.
Adverse events | 16 weeks
  Security of treatment (number of related adverse events in the two groups).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Gasperini, MD, Study Director — Medical Advisor
Locations (1):
- AOU Careggi - SOD Reumatologia - Scleroderma Unit, Florence, Italy

IPD SHARING:
Plan to Share IPD: No